CLINICAL TRIAL: NCT00115024
Title: Estrogen in the Prevention of Atherosclerosis Trial
Brief Title: EPAT: Estrogen in the Prevention of Atherosclerosis Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Mead Johnson Nutrition (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AG0026; R01AG018798 (NIH)
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2005-06

CONDITIONS: Atherosclerosis; Postmenopause
Keywords: cardiovascular disease; CVD; estrogen; cholesterol; LDL; lipids; postmenopausal
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

INTERVENTIONS:
Drug: Micronized 17B-estradiol

SUMMARY:
The purpose of this study is to determine the effects of estrogen replacement therapy (ERT) on the progression of early atherosclerosis in healthy postmenopausal women without preexisting cardiovascular disease (CVD).

DETAILED DESCRIPTION:
The primary goal of this randomized, controlled trial is to determine if ERT stabilizes, retards, and/or reverses the progression of atherosclerosis in postmenopausal women. We will further evaluate the association of lipid and non-lipid factors of ERT-mediated reduction in the progression of early atherosclerosis. Ultrasonography will be used to measure the rate of change in the thickness of the carotid artery. Blood samples will be used for measuring lipid and non-lipid mediators of ERT.

A total of 222 healthy postmenopausal women 46 to 80 years old without CVD symptoms will be randomized to receive either micronized 17B-estradiol (Estrace) 1mg/day, or a matching placebo tablet daily. All women will be on a low fat/low cholesterol diet, and will receive pravastatin if their LDL cholesterol level exceeds 160 mg/dL. Participants will undergo ultrasonography at baseline and every 6 months throughout the 2 years of randomized treatment. Measurements of lipid and non-lipid biochemical markers will also be done at baseline and every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female (serum estradiol less than 20 pg/ml)
* 46 to 80 years old
* Fasting LDL-C levels 130 to 210 mg/dL
* Triglyceride levels less than 400 mg/dL
* Current non-smoker

Exclusion Criteria:

* Clinical evidence of cardiovascular disease
* HDL-C level less than 30 mg/dL
* Fasting blood glucose greater than 200 mg/dL
* Previous hormonal replacement therapy (non-contraceptive) over 10 years duration and/or current use within 1 month
* Uncontrolled hypertension
* Untreated thyroid disease
* Renal insufficiency
* Clinical evidence of congestive heart failure
* Life threatening disease with prognosis less than 5 years
* Alcohol intake greater than 5 drinks per day (1 drink = 1 1/2 oz distilled spirits, 4 oz wine, or 12 oz beer) or substance abuse (intravenous drug abuse, cocaine use)
* History of estrogen dependent cancer or detected at screening or any other disorder precluding use of ERT
* Hot flashes greater than 5 per day which interfere with daily activity and preclude randomization to placebo.

Ages: 46 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222
Dates: Start 1994-04; Primary Completion 1998-11 (Actual); Study Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
rate of change of distal common carotid artery (CCA) far wall intima-media thickness (IMT)

SECONDARY OUTCOMES:
lipid and non-lipid factors

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, MD, Principal Investigator — University of Southern California, Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine
Locations (1):
- Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine, Los Angeles, California, United States

REFERENCES:
- [Result] Hodis HN, Mack WJ, Lobo RA, Shoupe D, Sevanian A, Mahrer PR, Selzer RH, Liu Cr CR, Liu Ch CH, Azen SP; Estrogen in the Prevention of Atherosclerosis Trial Research Group. Estrogen in the prevention of atherosclerosis. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2001 Dec 4;135(11):939-53. doi: 10.7326/0003-4819-135-11-200112040-00005. PMID 11730394
- [Derived] Steiner AZ, Xiang M, Mack WJ, Shoupe D, Felix JC, Lobo RA, Hodis HN. Unopposed estradiol therapy in postmenopausal women: results from two randomized trials. Obstet Gynecol. 2007 Mar;109(3):581-7. doi: 10.1097/01.AOG.0000251518.56369.eb. PMID 17329508